





# PROYECTO DE INVESTIGACION

## I. DATOS GENERALES.

1. Titulo del proyecto: Evaluación De La Eficacia De La N-Acetilcisteína Para Reducir El Craving Y Prolongar La Abstinencia De Pasta Base De Cocaína.

2. Patrocinador: Universidad de Concepción y

Fondo Nacional de Investigación y Desarrollo en Salud (FONIS).

3. Área de desarrollo: Investigación clínica

4. Duración: 2 años (2017 y 2018)

5. Investigadores

- Investigador responsable : Carmen Gloria Betancur Moreno.

Médico Psiquiatra.

PhD(c) en Salud Mental.

- Investigador alterno

: Benjamín de la Cruz Vicente Parada.

Médico Psiquiatra. PhD en Psiquiatría.

- Investigadores colaboradores:

Carolina Pilar Gómez Gaete, Co-Investigadora.

Químico Farmaceútico. PhD. En Farmacotecnia Biofarmacia. Rol en la Investigación: elaboración de los medicamentos. aleatorización de pacientes y supervisión del

María Paz Casanova Laudien. Co-Investigadora.

Estadístico. PhD en Estadística. Rol en la Investigación: Análisis de datos. Apoyo en metodología de la investigación y supervisión de la misma.

## II. DESCRIPCION DEL PROYECTO

# 1. ANTECEDENTES DE LA PROPUESTA:

#### 1.1. Planteamiento Del Problema

La Pasta Base de Cocaína (PBC) es una sustancia psicoactiva, fumable, obtenida al macerar las hojas de la planta erytroxilon coca con sustancias tales como el queroseno y el ácido sulfúrico, durante el primer paso del proceso de extracción de la cocaína 1,2. Tanto la mezcla con las sustancias antes mencionadas, como su vía de administración, le confieren a la PBC un gran poder adictivo y elevada toxicidad, ocasionando severos trastornos físicos, mentales y sociales a aquellos que la consumen<sup>3</sup>.







Chile se ha visto afectado por el consumo de esta sustancia desde fines de la década de los ochenta<sup>4</sup> llegando a ser, según el informe de la CICAD del año 2015<sup>5</sup>, el país latinoamericano con mayor prevalencia de consumo de esta sustancia en el último año en población escolar y el segundo con mayor prevalencia de consumo en población general. Por otra parte, al igual que en otros países del continente<sup>2</sup>, la clase social más pobre de nuestro país ha sido la más afectada con esta problemática<sup>6</sup>, con las ya mencionadas consecuencias sobre la salud física, mental y social de los individuos y su entorno, no existiendo a la fecha tratamientos con eficacia demostrada para ir en ayuda de aquellos que desean detener el consumo problemático de esta droga.

Uno de los grandes inconvenientes que existe para ofrecer un tratamiento eficaz a estos pacientes es que, dado que la PBC es una sustancia altamente adictiva, al ser retirada del organismo provoca un conjunto de síntomas de abstinencia, los cuales resultan tan molestos para los usuarios que regularmente deben volver a consumirla para aliviarse de ellos<sup>7</sup>. Uno de estos síntomas es el *craving*, el cual corresponde a un deseo intenso y urgente por consumir la sustancia una vez detenido su uso, con las consecuentes molestias físicas y psicológicas asociadas<sup>8</sup>. Este es, a su vez, uno de los síntomas más frecuentes de encontrar en quienes dependen de la PBC durante el período de abstinencia y se asocia regularmente a la recaída en el consumo de distintas drogas<sup>9</sup>. A la fecha no existen tratamientos aprobados por la *Food and Drug Administration* (FDA) en EEUU, así como tampoco por la Agencia Nacional de Medicamentos (ANAMED) del Instituto de Salud Pública (ISP) de Chile para el manejo del *craving* de cocaína, ni para el tratamiento de la dependencia de esta droga ni sus derivados, en ninguna de sus formas de uso<sup>10</sup>.

### 1.2 Justificación De La Investigación

El consumo de sustancias psicoactivas es un problema de salud pública a nivel mundial pues representa una importante carga de enfermedad para las naciones<sup>11</sup>. Según el último informe de la Organización de Naciones Unidas (ONU) del año 201512, se estima que un total de 246 millones de personas en el mundo (una de cada veinte personas de entre 15 y 64 años de edad), consumieron drogas ilícitas en 2013. Este mismo informe muestra que, si bien el consumo de estas sustancias se ha mantenido más o menos estable en los últimos cinco años, la magnitud del problema mundial de las drogas ha aumentado, pues las consecuencias de su consumo en la población han ido creciendo y con ello ha aumentado también la carga para los sistemas de salud pública en lo que respecta a prevención, tratamiento y rehabilitación de los trastornos relacionados con éstas. Esto se hace más evidente si se tiene en cuenta que más del 10% de los consumidores de drogas ilícitas en el mundo sufren trastornos ocasionados por el consumo de dichas sustancias y sólo uno de cada seis de estos consumidores problemáticos tiene acceso a tratamiento<sup>12</sup>. Por otra parte Degenhardt et al. 13 en su artículo sobre carga mundial de enfermedad atribuible al consumo y dependencia de drogas ilícitas en el mundo nos muestra que a nivel global los trastornos por consumo de drogas implicaron directamente casi 20 millones de años de vida perdidos







ZOIVITE ÉTICO

ajustados por discapacidad (AVAD) en 2010 lo que, a su vez, representa un 0,8% de todas las causas de AVAD en el mundo. Esa cifra supone además un incremento del 52% desde las estimaciones realizadas en el año 1990. Finalmente estos mismos autores comentan que si bien la principal carga de enfermedad está dada por los trastornos derivados del uso de opiáceos y derivados anfetamínicos, la cocaína sigue siendo la droga que mayor preocupación suscita en América Latina y el Caribe<sup>12,13</sup>.

Es en ese contexto, que resulta de gran preocupación el poder ofrecer una ayuda eficaz a aquellos pacientes que consultan por problemas derivados del consumo de cocaína y en particular en nuestro país en aquellos usuarios de una de sus formas fumables, la PBC. Según el Décimo Primer Estudio Nacional de Drogas en Población General en Chile publicado por el Servicio Nacional Para la Prevención y Rehabilitación de Drogas y Alcohol (SENDA) el año 2015<sup>6</sup>, la prevalencia de último año de consumo de PBC alcanza al 0,5% de la población general, lo que representa un leve aumento en la prevalencia con respecto al mismo estudio del año 2012. En este mismo estudio se detecta además un aumento significativo del consumo de PBC en la clase socioeconómica más baja del país, así como en el grupo etario de 35 a 44 años. Por otra parte, según el Informe Semestral 2015 del Área de Tratamiento y Rehabilitación del SENDA<sup>14</sup>, el 39,9% de los usuarios de los diferentes servicios de atención para drogodependientes en Chile tienen a la PBC como droga principal de consumo, siendo este porcentaje aún mayor entre las mujeres (42,2% de las usuarias), superando la tasa de consultantes por trastornos por consumo de Alcohol (38,1%) y muy por encima de la de aquellos con trastorno por uso de Clorhidrato de Cocaína (15,3%) y de Marihuana (5%).

Ahora bien, el principal problema de la PBC no es su prevalencia en la población chilena, sino la carga de enfermedad que representa para nuestro país dado todos problemas sanitarios y sociales derivados de su consumo. Entre ellos está el trastorno mental conocido como dependencia o trastorno por consumo moderado a grave, según la quinta versión del Manual Diagnóstico y Estadístico de la Asociación Americana de Psiquiatría (DSM-V)<sup>15</sup>. Según el último estudio del SENDA en población general<sup>6</sup>, la PBC es la droga que presenta mayor tasa de dependencia entre quienes la consumen con una prevalencia de ésta de 65,6% entre los consumidores del último año.

Por otra parte quienes tienen consumo problemático de cocaína y sus drivados (lo que incluye a la PBC) suelen tener una alta tasa de comorbilidad tanto psiquiátrica como médica asociada, al igual que la mayoría de los pacientes con trastorno por consumo de sustancias <sup>16-22</sup>. Dentro de la comorbilidad psiquiátrica destacan los trastornos del estado de ánimo (26,6%) y los trastornos de ansiedad (13%)<sup>22</sup>. Respecto de la comorbilidad médica, es amplia la literatura en torno a las consecuencias tanto del uso agudo como crónico de la cocaína y sus derivados, destacando en ella la evidencia contundente acerca del daño pulmonar secundario al uso de cocaína fumada<sup>23-29</sup>, así como de otras complicaciones médicas asociadas al consumo de esa y otras formas de cocaína. Ahora, respecto de otros riesgos sobre la salud, Santis et al<sup>30</sup> encuentran en su estudio sobre consumidores de PBC no consultantes en Chile, que éstos presentan una mayor proporción de conductas de riesgo en







la vida, de tipo sexual (nunca uso de anticoncepción, sexo por dinero y droga por sexo), autolesiones, intento de suicidio, además de negligencia en el cuidado de menores, comisión de delitos y porte de armas, entre otros. Finalmente, y ligado con este último punto, no se pueden desconocer las consecuencias que el consumo problemático de PBC ha tenido sobre la seguridad pública en los últimos años en Chile, pues tal como lo describen Valenzuela y Larroulet<sup>31</sup> en su texto sobre la relación droga y delito, el consumo de PBC se ha visto relacionado regularmente con la violencia en barrios donde la distribución y venta de esta sustancia, unida a situaciones de vulnerabilidad social y económica, constituye la base para la articulación de grupos criminales ligados al narcotráfico.

El asunto aquí es que, pese a la fuerza de los datos enunciados en este apartado, en los que se destaca la carga sanitaria y social que representa el consumo problemático de cocaína y sus derivados, entre los que se incluye la PBC, sólo el 4,5% de los individuos con consumo riesgoso de drogas ilícitas, recibe algún tipo de tratamiento<sup>32</sup>, no teniendo además a la fecha un protocolo de tratamiento estandarizado y eficaz para ayudar a los pacientes con trastorno por consumo de PBC a aliviar sus síntomas de abstinencia y con ello a la vez prolongar su tiempo sin consumir dicha sustancia.

Es en ese contexto que se justifica plantear este proyecto de investigación clínica, como un intento por sistematizar la observación e intervención inicial en los pacientes con trastorno por consumo de PBC en Chile, intentando al mismo tiempo encontrar un tratamiento eficaz para el manejo de los síntomas de abstinencia de dichos pacientes, en particular para el manejo del *craving* de PBC, el cual, como ya se ha dicho, es uno de los síntomas más constantes en pacientes que intentan detener su consumo. En la búsqueda, entonces, de ayudar a estos pacientes a aliviar dicho síntoma, y de esa forma también ayudarles a prolongar la abstinencia de esta sustancia, se encuentran en la literatura algunos trabajos recientes que apuntan a modificar la neurotransmisión glutamatérgica<sup>34-36</sup> en pacientes con dependencia de cocaína, en particular a través de la utilización de la N-Acetilcisteína (NAC) <sup>37-44</sup>.

En Chile la NAC es utilizada desde hace ya varios años con otros fines terapéuticos 45-46, tales como el tratamiento de las afecciones bronquiales agudas y crónicas, de la enfermedad pulmonar obstructiva crónica (EPOC), de la fibrosis quística, de la intoxicación por paracetamol y como protector renal o hepático, entre otros 46-47, siendo a la vez un medicamento muy seguro de utilizar. Es en ese contexto, y apoyándose en los antecedentes previamente expuestos, que se plantea este proyecto de investigación clínica en el cual se administraría NAC a pacientes con trastorno por consumo de PBC de modo de evaluar si la utilización de dicho fármaco en ellos les ayuda a reducir el *craving* por esta sustancia y así les permite prolongar el tiempo de abstinencia de la misma, con la consecuente reducción de riesgo de comorbilidad médica, psiquiátrica y "social", ya comentada. Finalmente es importante destacar que llevar a cabo este proyecto nos permitiría, además, establecer una base de trabajo para el desarrollo de una línea de investigación clínica en población usuaria.







de ésta y otras sustancias psicoactivas realizando de ese modo un aporte al desarrollo de la salud pública nacional.

#### 2. OBJETIVOS DEL PROYECTO Y SUPUESTO DE INVESTIGACIÓN:

#### 2.1. PREGUNTA DE INVESTIGACIÓN

¿Es la N-Acetilcisteína (NAC) capaz de reducir el el craving por Pasta Base de Cocaína (PBC) y ayudar a prolongar el tiempo de abstinencia de la misma, en pacientes con trastorno por consumo de esta sustancia?

#### 2.2. HIPÓTESIS DE INVESTIGACIÓN

H1: La NAC reduce el *craving* y ayuda a prolongar el tiempo de abstinencia de PBC, en pacientes con trastorno por consumo de esta sustancia.

#### 2.3. OBJETIVOS:

Objetivo General: Evaluar el efecto que tiene la NAC sobre el *craving* de PBC y la duración de la abstinencia de la misma, en pacientes con trastorno por consumo de esta sustancia.

#### **Objetivos Específicos:**

- 1. Evaluar el efecto de la NAC sobre el craving de PBC en usuarios con trastorno por consumo de esta sustancia.
- 2. Evaluar el efecto que tiene la NAC sobre la duración de la abstinencia de PBC en pacientes con trastorno por consumo de la misma.
- 3. Evaluar el efecto de la NAC sobre la tasa de caídas en el consumo de PBC en pacientes con trastorno por consumo de dicha sustancia.

#### 3. ESTADO DEL ARTE:

# 3.1. Adicción A La Cocaína Y Su Relación Con La Neurotransmisión Glutamatérgica:

Los efectos reforzantes y, por lo tanto, el alto potencial adictivo de la cocaína se han explicado fundamentalmente por su capacidad de activar los tractos mesolímbicos y/o mesocorticales dopaminérgicos, particularmente a nivel del núcleo accumbens<sup>48</sup>. De hecho, la potenciación de la neurotransmisión dopaminérgica es considerada habitualmente como el neurotransmisor más importante en la producción de los efectos subjetivos de la cocaína, así como de la inducción de las conductas estereotipadas y la estimulación de la actividad locomotora<sup>49</sup>. Sin embargo, la compleja interacción con otros sistemas de neurotransmisión es esencial para entender la intensa euforia y las propiedades reforzantes de la cocaína, así como el fuerte *craving* que se genera al dejar de consumirla.

Hoy sabemos que la neuromodulación glutamatérgica en el núcleo accumbens ejerce un papel esencial en los procesos que desencadenan la aparición del *craving*, las recaídas y el mantenimiento de la adicción<sup>50-52</sup>. De hecho, a través de diferentes mecanismos, la Versión 2. Fecha: 20 de marzo de 2017







neurotransmisión glutamatérgica está implicada en las conductas relacionadas con las búsquedas de las distintas drogas de abuso y los recuerdos asociados con el uso de éstas. Además, por lo general, la atenuación de la transmisión glutamatérgica reduce el refuerzo, la recompensa y las conductas asociadas con las recaídas a las diversas sustancias, mientras que la potenciación de la transmisión glutamatérgica parece facilitar las conductas de búsqueda de drogas. El papel de las vías glutamatérgicas en los efectos reforzantes y de recompensa y, por lo tanto en el potencial adictivo de la cocaína, ha sido claramente demostrado mediante estudios farmacológicos con antagonistas de los receptores glutamatérgicos<sup>53</sup>. De este modo, se sabe que los efectos del glutamato a nivel del núcleo accumbens jugarían un papel predominante como precipitante de una recaída en un sujeto dependiente de cocaína, habiéndose incluso sugerido que el glutamato sería más esencial para la adicción a la cocaína que la dopamina una vez establecida dicha adicción<sup>50</sup>.

# 3.2 Fármacos Con Acción Glutamatérgica En El Tratamiento De La Adicción A La Cocaína

A la fecha han sido múltiples los fármacos que se han utilizado en el tratamiento de la dependencia de cocaína, los cuales además han apuntado a una acción sobre distintos niveles de la neurotransmisión cerebral. Sin embargo en los últimos quince años aproximadamente, parte importante de la atención en torno a este tema se ha centrado en los agentes farmacológicos que modulan la neurotransmisión glutamatérgica, los cuales en algunas ocasiones han mostrado un resultado muy prometedor en el abordaje de la adicción a la cocaína. Entre estos agentes se encuentra un pro-fármaco de la cisteína conocido como N-Acetil-Cisteína (NAC).

#### 3.2.1. N- Acetilcisteína (NAC)

La NAC es un derivado del aminoácido cisteína utilizado habitualmente como mucolítico con múltiples mecanismos de acción, incluyendo el aumento de la síntesis de glutatión. Dado que la NAC es un pro-fármaco de la cistina, puede actuar como un substrato del intercambiador cistina-glutamato, que facilita el intercambio de moléculas de cistina extracelular por glutamato intracelular en la glía, y a su vez aumenta los niveles de glutamato extracelular en muchos tejidos, inclusive a nivel cerebral<sup>54</sup>. Específicamente, se ha hipotetizado que la NAC equilibraría y restablecería los niveles de glutamato extracelular en determinadas regiones como el núcleo accumbens, que si bien aumentan durante la exposición aguda a la cocaína sufren una depleción tras la abstinencia de la exposición repetida, posiblemente por la desensibilización de los autorreceptores presinápticos mGluR del Grupo II. Con la "normalización" de los niveles de glutamato extracelular en el circuito de recompensa se prevendría la liberación de glutamato con nuevas dosis de cocaína y la conducta de búsqueda de droga<sup>53,54</sup>. En un estudio cruzado, doble ciego, controlado con placebo se observó una inhibición del craving de cocaína inducido por estímulos, asociado con el tratamiento con NAC en dosis de 1.200 mg diarios<sup>40</sup>, sugiriéndose por lo tanto esta opción farmacológica para el abordaje de pacientes dependientes de cocaína. De hecho, Versión 2. Fecha: 20 de marzo de 2017









sendos estudios abiertos no sólo han mostrado la buena tolerabilidad de la NAC y la tendencia a la reducción del craving de cocaína<sup>37</sup>, sino que, además, en el segundo de ellos, un estudio de cuatro semanas de seguimiento, con dosis entre 1.200 y 3600 mg/día de NAC, la administración de este fármaco se asociaba con reducciones significativas en el consumo de cocaína<sup>38</sup>.

# 3.3. Abordaje Del Paciente Con Trastorno Por Consumo De PBC:

## 3.3.1. Evaluación Clínica: Instrumentos De Evaluación Del Síndrome De Abstinencia De PBC:

No existen instrumentos diseñados para evaluar el craving de PBC. Lo único que tenemos hoy son algunos instrumentos conocidos para evaluar el craving de cocaína, los cuales son de distintos tipos<sup>55</sup>. Inicialmente se utilizaron escalas unidimensionales de tipo analógico visual, en las que se pregunta al sujeto directamente por su deseo de consumir, situando en uno de los extremos de la línea la "ausencia de deseo" y en el otro el "deseo muy intenso". Entre estas escalas destacan la Cocaine Craving Scale56, la Minnesota Cocaine Craving Scale<sup>57</sup> y, más recientemente, la Escala Analógico Visual del Craving (EVA-Craving), diseñada y validada en español por Iraugi Castillo58.

Entre las escalas más amplias, tipo likert por ejemplo, destaca el Cocaine Craving Questionnaire (CCQ) desarrollado por Tiffany y cols. 59 que, como señalan Tejero, Trujols y Siñol<sup>60</sup>, el cual evalúa deseo de consumir cocaína, intención y planificación del consumo de cocaína, anticipación de los efectos positivos del consumo, anticipación de una mejora de los síntomas de abstinencia y pérdida de control sobre el consumo. Es un cuestionario autoadministrado y consta de 45 ítems, a los que el paciente debe de responder en una escala tipo Likert que va de cero a siete, en donde el cero representa muy en desacuerdo y el siete muy de acuerdo. La evaluación se centra en el momento presente o en los últimos siete días, siendo un instrumento con validez y fiabilidad satisfactorias que, mediante análisis factorial, confirma la estructura multidimensional del craving<sup>62</sup>. En cuanto a las limitaciones de este cuestionario está su extensión, lo que dificulta su utilización en investigaciones en las que el craving sea una variable más a medir, existiendo entonces una versión abreviada llamada CCQ-N-10, validada al espeñol por Iraurgi Castillo y cols. 58, la cual consta de 10 ítems y evalúa los síntomas de craving al momento de la entrevista.

Finalmente, para evaluar más ampliamente el síndrome de abstinencia de cocaína, privilegiando al mismo tiempo el uso de cuestionarios breves, se ha diseñado la Escala de Valoración de la Gravedad Selectiva para Cocaína (CSSA), la cual fue creada por Kampman y cols<sup>61</sup> a fines de los años noventa y consiste en una entrevista semi-estructurada, heteroaplicada, de 18 ítems en los que se evalúan signos y síntomas que se han asociado con más frecuencia a la abstinencia inicial de cocaína. Cada signo y síntoma se evalúa mediante una escala de intensidad o frecuencia de 8 puntos que van de 0 a 7, donde 0 es ausente y 7 es la máxima intensidad o frecuencia de cada signo o síntoma. El rango de puntuaciones oscila Versión 2. Fecha: 20 de marzo de 2017







entre 0 y 126, no teniendo un puntaje de corte establecido, sino que a mayor puntuación mayor gravedad de la abstinencia de cocaína, permitiendo hacer un seguimiento en el tiempo a los pacientes para evaluar su evolución. Este cuestionario fue adaptado y validado al español hace un par de años por Pérez de los Cobos y su equipo<sup>62</sup>, siendo utilizado y citado en diversas investigaciones recientes que miden *craving* y/o síntomas de abstinencia inicial de cocaína <sup>38,39,63,64</sup>.

Por todo lo anteriormente expuesto es que en esta investigación se ha privilegiado utilizar el EVA-craving, el CCQ-N-10 y el CSSA, para medir el craving y los síntomas de abstinencia de PBC en los pacientes ingresados al estudio.

# 3.3.2. Tratamientos Actuales Para Los Trastornos Por Uso De PBC

A la fecha no existen tratamientos específicos para el manejo de los trastornos por consumo de PBC en el mundo. Por otra parte, tal como se ha mencionado previamente, no existen tampoco tratamientos farmacológicos aprobados por la FDA en los EEUU ni por ANAMED en Chile, para el manejo de los trastornos por consumo de cocaína y sus derivados, habiéndose intentado a la fecha múltiples aproximaciones terapéuticas, sin resultados sólidos que nos permitan generar protocolos claros de intervención para estos pacientes.

En Chile, los tratamientos existentes actualmente para pacientes con trastornos por uso de PBC y otras drogas son diseñados y regulados por el SENDA, organismo que contempla tres planes de intervención diferenciados de acuerdo a la complejidad diagnóstica de los pacientes<sup>33</sup>. Estos planes son: de tipo residencial, de tipo ambulatorio intensivo y de tipo ambulatorio básico, los que, a su vez, son ejecutados por un equipo multidisciplinario capacitado y con competencias clínicas (médico, psicólogo, asistente social, psiquiatra, técnico en rehabilitación, terapeuta ocupacional, enfermera) en establecimientos de salud públicos o en centros de tratamiento privados autorizados por la SEREMI de Salud crrespondiente y que están en convenio con el SENDA. Este equipo realiza actividades terapéuticas individuales, familiares, grupales y comunitarias (incluyendo consulta médica, psiquiátrica, de salud mental y psicológica, psicodiagnóstico, intervención psicosocial de grupo, visita domiciliaria, exámenes y fármacos).

Ahora bien, pese a que existe una normativa vigente<sup>65-67</sup> para planificar las intervenciones antes mencionadas, de acuerdo a la complejidad de los pacientes, no existe a la fecha un protocolo de tratamiento farmacológico estandarizado y eficaz para ayudar a los pacientes con trastorno por consumo de PBC a aliviar sus síntomas de abstinencia y con ello a la vez prolongar su tiempo sin consumir dicha sustancia.

## 4. METODOLOGIA (DISEÑO DEL PROYECTO)

A. CLASIFICACIÓN: cuantitativa

B. TIPO DE ESTUDIO: Se trata de un estudio experimental, correspondiente a un ensayo clínico aleatorizado, doble ciego, controlado, de fase II, en el cual se evaluará la Versión 2. Fecha: 20 de marzo de 2017







utilidad clínica de la n-acetileisteína (NAC) para el manejo del síndrome de abstinencia de pasta base de cocaína (PBC). Es un estudio de tipo explicativo, con diseño de grupos paralelos.

#### C. VARIABLES:

C.1. Variables de resultado primarias: las principales variables de resultado serán la reducción del craving de PBC y la duración de la abstinencia de la misma. Lo primero se medirá con escala de Escala Visual Análoga (EVA-Craving), cuyos valores de medición van desde el 0 al 100, donde 0 representa "sin craving o deseo de consumo por PBC" y 100 representa el "máximo deseo o craving por consumir la PBC". En paralelo a la utilización de la EVA-Craving, se utilizará el Cocaine Craving Questionnaire-Now (CCQ-N-10), específico para cocaína y adaptado para PBC, además de la Escala de Valoración de la Gravedad Selectiva para Cocaína (CSSA) para medir sintomatología de abstinencia de cocaína (PBC). Lo segundo se medirá llevando un registro de los días de abstinencia de PBC desde el ingreso al estudio hasta las fechas de las distintas evaluaciones.

C.2. Variable de resultado secundaria: será la tasa de caídas en el consumo de PBC de los pacientes de ambos grupos de tratamiento, lo cual se objetivará contando el número de pacientes que caen en el consumo de PBC durante el mes de tratamiento y la proporción de éstos en cada grupo.

## C.3. Posibles variables intervinientes:

- Predisposición de los pacientes con respecto al tratamiento: se controlará al no informar o hacer "ciegos" a los pacientes respecto de cuál será el tratamiento recibido.
- Efecto inductor del terapeuta sobre el paciente: se controlará al "hacer ciego" al tratamiento indicado también al médico tratante.
- Efecto de otras drogas: relativamente controlada al exigir, como criterio de ingreso al
  estudio, la PBC como droga principal de consumo.
- Efecto de otros tratamientos: se controlará al realizar el estudio sin la aplicación de otros fármacos para tratamiento de adicciones ni psicoterapia, ya que el estudio se realizará en un tiempo breve, transcurriendo un máximo de 28 días entre el inicio y el fin del tratamiento. En este punto es importante aclarar que, si bien no se usará otro tratamiento farmacológico estándar para el manejo de los síntomas de abstinencia de PBC (dado que no existe), en caso de que el paciente se encuentre en tratamiento previamente con algún agente farmacológico por otros síntomas (ej., inductor del sueño por insomnio o antipsicótico por trastorno conductual), este tratamiento se mantendrá durante el estudio. Del mismo modo, en caso de que el paciente manifieste angustia intensa u otro síntoma que desajuste su conducta de modo importante durante el estudio, se usará farmacoterapia estándar en dichos casos. A saber:

O Quetiapina entre 25 y 100 mg en caso de crisis de angustia o insomnio pertinaz.









- Quetiapina entre 100 mg/d y 200 mg/d en caso de descontrol de impulsos o desajuste conductual agudo (riesgo agitación).
- Sesgo respecto de la intencionalidad de participar o no en el estudio: controlado dado que todos quienes ingresen lo harán voluntariamente y firmarán un consentimiento donde quede explicitado aquello.
- Sesgo al elegir los pacientes de cada grupo: controlado gracias a la aleatorización de los pacientes, la cual se realizará de la siguiente forma:
  - o Los pacientes serán aleatorizados en dos grupos, los cuales se llamarán Grupo I y Grupo II y será distribuidos en ellos de acuerdo a un sistema de aleatorización por bloques, realizado por la farmacóloga que apoyará a la investigadora en la investigación. Será ella quien sorteará los pacientes a incorporar en cada grupo, cada 10 pacientes que sean reclutados, poniendo todos los números de ese grupo de pacientes en una tómbola y número por medio se asignará un paciente al mismo grupo. Con ello la farmacóloga generará una tabla con los pacientes pertenecientes a ambos grupos, en cada bloque, y la investigadora será ciega a esto manejando los sobres con los fármacos a entregar con sus respectivos números sin saber a qué grupo corresponde cada uno.

#### D. POBLACION:

Pacientes con trastorno por consumo de pasta base de cocaína (PBC) consultantes de centros de atención ambulatoria en salud mental del Servicio de Salud Concepción durante los años 2017 y 2018.

#### E. MUESTRA:

La muestra estará compuesta por 106 (ciento seis) pacientes con trastorno por consumo de PBC (53 por cada brazo), consultantes de centros de atención ambulatoria en salud mental del Servicio de Salud Concepción (COSAM Concepción, CT. Anün, COSAM Lota y Servicio de Psiquiatría del HCRC). El tamaño de la muestra se ha calculado en relación al tamaño del efecto (TE) de la NAC, encontrado en estudios previos en que se ha tratado a pacientes dependientes de cocaína con este fármaco, para reducir el craving y/o prolongar la abstinencia de esta sustancia. La muestra, entonces, tendrá suficiente poder estadístico (β=0.8) para detectar al menos un TE del tratamiento de d=0,55 (calculado con los datos de estudios previos con este fármaco en pacientes dependientes de cocaína<sup>37</sup>) y considerando que el análisis de resultados se hará mediante una prueba más poderosa que tpara muestras independientes, aceptando un nivel de significación α= 0,05, en un diseño de dos colas. Es importante destacar que, dadas las características de estos pacientes, se espera que aproximadamente un 40% de aquellos ingresados al estudio deserten de éste, por lo que en la aleatorización y asignación de pacientes a tratamiento deberán considerarse al menos 148 participantes. Por otro lado, se estima aproximadamente un 50% de pérdida tras el enrolamiento debido a los criterios de exclusión y a la no aceptación de participación por







parte de algunos de ellos, por lo que probablemente se tendrá que entrevistar a un mínimo de 300 pacientes.

#### Criterios de inclusión:

- Ser paciente de alguno de los centros de atención participantes del estudio o estar en busca de tratamiento en alguno de dichos centros.
- Tener 18 años de edad o más.
- Cumplir con los criterios de trastorno por consumo de cocaína (PBC) de acuerdo al DSM-V (Por lo tanto debe tener al menos un año de consumo de esta sustancia).
- Tener a la PBC como droga principal de consumo.
- Haber consumido PBC en el mes previo al inicio del tratamiento.
- Tener historia de algún síntoma de abstinencia de PBC previo o al momento del ingreso al estudio.
- Aceptar participar de este estudio y firmar consentimiento informado para ingresar al mismo.

#### Criterios de exclusión:

- Estar embarazada o amamantando.
- Tener dependencia de alguna otra sustancia distinta de PBC, alcohol, nicotina o marihuana.
- Presentar un síndrome de abstinencia severo de alcohol durante el estudio.
- Estar cursando un delirium al momento del estudio.
- Tener algún trastorno psiquiátrico que disminuya su capacidad de consentir y/o participar adecuadamente del estudio (retardo mental, trastorno psicótico, trastorno generalizado del desarrollo u otro de esa naturaleza).
- Tener diagnóstico de úlcera péptica.
- Tener diagnóstico de asma bronquial o enfermedad respiratoria grave.
- Tener epilepsia o historia de convulsiones.
- Tener alguna enfermedad médica grave conocida y/o en tratamiento (ej. cáncer, insuficiencia hepática o renal).
- Estar utilizando al momento del estudio fármacos como penicilina, tetraciclina, carbamazepina, nitroglicerina, antitusivos o inhibidores de la secreción bronquial.
- Tener antecedente de alergia a la NAC.

## F.INSTRUMENTOS DE RECOLECCION DE DATOS:

#### F.1. Para La Valoración Clínica Inicial Del Paciente:

a. Entrevista semi-estructurada: diseñada específicamente para esta investigación. Se aplicará, al momento de su ingreso, a todos los pacientes que lleguen a consultar al centro de atención clínica donde se esté desarrollando la investigación y que tengan como motivo de consulta un consumo problemático de PBC. Será un psiquiatra quien la aplique y en ella se recogerán datos socio-demográficos de los pacientes, tales







como sexo, edad, estado civil, escolaridad, entre otros. Además en ella se recogerán datos respecto del consumo de PBC y de otras drogas, entre los que se incluirá edad del primer consumo, edad de inicio del consumo regular (entendiéndose éste como consumo al menos una vez al mes), frecuencia del consumo en el último año, dosis utilizada regularmente en el último año, fecha del último consumo, tiempo máximo sin consumo tras el inicio del uso regular de la droga, síntomas de abstinencia experimentados al cesar el consumo, período de máximo uso de la droga en su vida y dosis usada en ese período, entre otros. Se adjunta esta entrevista en los anexos de este proyecto.

b. Entrevista Neuropsiquiátrica Internacional (MINI): También será aplicada por un psiquiatra al momento del ingreso de los pacientes al centro de atención ambulatoria, para obtener información estandarizada respecto de otros posibles diagnósticos psiquiátricos que pudiesen excluir a los pacientes del estudio. Esta consiste en una entrevista diagnóstica estructurada de breve duración que explora los principales trastornos psiquiátricos del Eje I del DSM-IV y la CIE-10. Estudios de validez y de confiabilidad se han realizado comparando la MINI con el SCID-P para el DSM-III-R y el CIDI (una entrevista estructurada desarrollada por la Organización Mundial de la Salud para entrevistadores no clínicos para la CIE-10). Los resultados de estos estudios demuestran que la MINI tiene una puntuación de validez y confiabilidad aceptablemente alta, pero puede ser administrada en un período de tiempo mucho más breve (promedio de  $18,7 \pm 11,6$  minutos, media 15 minutos) que los instrumentos mencionados. Puede ser utilizada por clínicos tras una breve sesión de entrenamiento. Entrevistadores no clínicos deben recibir un entrenamiento más intenso<sup>68,69</sup>

# F.2. Para La Evaluación De La Gravedad Del Cuadro Clínico Y De Su Evolución:

Escala de Impresión Clínica Global (ICG): es una escala descriptiva que proporciona información cualitativa acerca de la gravedad del cuadro clínico y de su evolución<sup>69</sup>. Consta de dos sub-escalas: la primera para medir gravedad del cuadro clínico y la segunda para evaluar la mejoría del cuadro en relación a las intervenciones terapéuticas. Amabas sub-escalas constan de un único ítem de 8 puntos con rango de 0 a 7, siendo las especificaciones de cada nivel para la primera sub-escala, las siguientes: 0= no determinado; 1-2= no del todo enfermo o dudosamente enfermo; 3= ligeramente enfermo, 4= moderadamente enfermo; 5= gravemente enfermo; 6= severamente enfermo y 7= grado más extremo de la enfermedad. En el caso de la segunda sub-escala, la valoración también va de 0 a 7, tal como se describe a continuación: 0= No evaluado; 1= Mucho mejor; 2= Moderadamente mejor; 3= Levemente mejor; 4= Sin cambios; 5= Levemente peor; 6= Moderadamente peor y 7= Mucho peor. Se aplicará al inicio del tratamiento, a las 2 y a las 4 semanas de tratamiento.

F.3. Para La Valoración Clínica Del Cumplimiento Terapéutico:

Test de Morisky-Green: Este método, que está validado para diversas enfermedades









COMMITE

crónicas, fue desarrollado originalmente por Morisky, Green y Levine<sup>70</sup> para valorar el cumplimiento de la medicación en pacientes con hipertensión arterial (HTA). Desde que el test fue introducido se ha usado en la valoración del cumplimiento terapéutico en diferentes enfermedades. Consiste en una serie de 4 preguntas de contraste con respuesta dicotómica sí/no, que refleja la conducta del enfermo respecto al cumplimiento. Se pretende valorar si el enfermo adopta actitudes correctas con relación con el tratamiento para su enfermedad; se asume que si las actitudes son incorrectas el paciente es incumplidor. Presenta la ventaja de que proporciona información sobre las causas del incumplimiento. Las preguntas, que se deben realizar entremezcladas con la conversación y de forma cordial, son las siguientes:

- 1. ¿Olvida alguna vez tomar los medicamentos para tratar su enfermedad?
- 2. ¿Toma los medicamentos a las horas indicadas?
- 3. Cuando se encuentra bien, ¿deja de tomar la medicación?
- 4. Si alguna vez le sienta mal, ¿deja usted de tomarla?

El paciente es considerado como cumplidor si se responde de forma correcta a las 4 preguntas, es decir, No/Si/No/No.

### F.4. Para La Valoración Clínica De la Abstinencia:

- a. Evaluación de los Días de Abstinencia de PBC: se medirá tanto por el reporte del paciente como a través de la aplicación de test de drogas en orina para corroborar esta información.
- b. <u>Evaluación de los Síntomas de Abstinencia:</u> Se evaluará registrando en la entrevista clínica los síntomas referidos por el paciente, así como también por la aplicación del siguiente instrumento:

Escala de Valoración de la Gravedad Selectiva para Cocaína (Cocaine Selective Severity Assessment, CSSA): Es una entrevista semi-estructurada, hetero-aplicada, de 18 ítems en los que se evalúan signos y síntomas que se han asociado con más frecuencia a la abstinencia inicial de cocaína. Cada signo y síntoma se evalúa mediante una escala de intensidad o frecuencia de 8 puntos que van de 0 a 7, donde 0 es ausente y 7 es la máxima intensidad o frecuencia de cada signo o síntoma. El rango de puntuaciones oscila entre 0 y 126, no teniendo un puntaje de corte establecido, sino que a mayor puntuación mayor gravedad de la abstinencia de cocaína, permitiendo hacer un seguimiento en el tiempo a los pacientes para evaluar la evolución tanto del craving de cocaína como de otros síntomas de abstinencia de dicha sustancia. Este cuestionario fue adaptado y validado al español hace un par de años por Pérez de los Cobos y cols<sup>62</sup>, mostrando en dicho proceso de validación una adecuada consistencia interna global, con un coeficientes alfa de Cronbach de 0,84, sacando la bradicardia y considerando los restantes 17 ítems como un único constructo, sin embargo detectó en dicho proceso de validación algunos ítems problemáticos como los de hiperfagia, hipofagia, bradicardia y síntomas.







depresivos. Por otra parte la matriz de correlación para el modelado de análisis factorial fue alta, ya que la medida del KMO fue de 0,777 y la prueba de esfericidad de Bartlett fue estadísticamente significativa (p=0,001) y la fiabilidad test-retest medida a través de la ICC produjo un excelente valor de 0,87 (IC del 95%: 0,82 a 0,90) al considerar el test sin el ítem de bradicardia incluido.

# F.5. Para La Valoración Clínica Del Craving:

- a. Escala Analógico Visual del Craving (EVA-Craving): Es una escala analógico visual de 100 milímetros basada en la Escala de Craving a Cocaína de Voris, diseñada y utilizada por Iraugi Castillo y colaboradores en el proceso de validación del CCQ-N-10 al español<sup>58</sup>, para valorar "el deseo o ganas de consumir durante las últimas 24 horas". En dicho proceso de validación se presentaba al entrevistado esta escala graduada a modo de termómetro situándose en el extremo inferior o izquierdo el lema "ningún deseo" y en el extremo superior o derecho el lema "Incapaz de resistirme"; debiendo señalar con una raya aquel punto de la escala que representase su valoración del grado de deseo percibido. El resultado es una puntuación de escala continua entre 0 y 100 tomándose como valor la distancia medida con regla entre el extremo inferior o izquierdo y el punto de señalado por el entrevistado. Sirve, en este caso, básicamente para ver variaciones intra-sujeto del deseo, ansias o craving de consumo de cocaína.
- b. Cuestionario de Craving de Cocaína (Cocaine Craving Questionnaire-Now, CCQ-N-10): Cuestionario auto-administrado, de 10 ítems tipo Likert cuyos puntajes van de 1 a 7, los cuales se centran en el craving por cocaína en el momento presente. En su versión y adaptación en español de este instrumento<sup>58</sup> el alpha de Cronbach alcanzó un valor de 0,947 mostrando con ello una adecuada consistencia interna. La fiabilidad test-retest proporcionó un valor de correlación de Pearson de 0,61 y un Coeficiente de Correlación Intraclase (ICC) de 0,59. Por otro lado, y anticipándonos a los resultados del análisis factorial confirmatorio, a partir de los coeficientes Lambda-X y Theta-Delta se obtuvo una fiabilidad de constructo de 0,948 con un porcentaje de varianza extractada del 65,3%. El Análisis Factorial Exploratorio (AFE) presentó valores óptimos para las pruebas de Kaiser-Meyer-Olkin (KMO), siendo ésta de 0,85 y de esfericidad de Bartlett (622,5; p< 0,001), obteniéndose un único factor que explicó una varianza total del 68,6%, con pesos factoriales por encima del valor 0,70 en todos los casos salvo para el ítem 8 que alcanzó un valor de 0,64. Por otro lado el Análisis Factorial Confirmatorio (AFC) mostró pesos factoriales altos en general, salvo en el caso del ítem 8

#### G. PROCEDIMIENTO:

 a. <u>Selección de los Pacientes:</u> un psiquiatra realizará una evaluación clínica a todos los pacientes que lleguen a los centros de atención ambulatoria participantes y que Versión 2. Fecha: 20 de marzo de 2017

> CIENT CIENT





refieran como motivo de consulta principal "un consumo problemático de PBC". Dicha evaluación será realizada utilizando la entrevista semi-estructurada diseñada para este estudio y la *Mini-International Neuropsychiatric Interview* (MINI), con las cuales se detectará si el paciente cumple con los criterios de inclusión y si no presenta algún criterio de exclusión para esta investigación. Una vez seleccionado cada potencial participante, se le invitará a participar del estudio, explicándole la naturaleza de éste, solicitándole posteriormente que lea y firme un consentimiento informado, en caso de aceptar participar en él. Ingresarán al estudio, entonces, sólo aquellos pacientes que, cumpliendo con los criterios de selección, hayan firmado el consentimiento informado correspondiente.

- b. <u>Tratamientos a Administrar</u>: En este estudio se administrará uno de los siguientes tratamientos a los pacientes participantes de él:
  - Tratamiento con N- Acetilcisteína (NAC): consistente en la administración por vía oral de 2 cáspulas que contengan 600 mg de este fármaco cada una, cada 12 hrs.
  - O Tratamiento con Placebo: consistente en la administración por vía oral, también cada 12 hrs, de 2 cápsulas iguales a las de NAC en tamaño, forma y color, pero que contengan una sustancia sin acción farmacológica, denominada placebo.
- c. Asignación a los Grupos de Tratamiento: Tras su ingreso al estudio, los pacientes se asignarán aleatoriamente a uno de los dos grupos de tratamiento, según la tabla generada previamente por la farmacóloga del equipo investigador de acuerdo a un sistema de aleatorización por bloques. Dicha aleatorización, descrita previamente, se realizará sorteando a los pacientes a incorporar en cada grupo, cada 10 pacientes que sean reclutados, poniendo todos los números de ese grupo de pacientes en una tómbola y número por medio se asignará un paciente al mismo grupo. Con ello la farmacóloga generará una tabla con los pacientes pertenecientes a ambos grupos, en cada bloque, y numerará los sobres con los diferentes tratamientos a administrar de acuerdo a ello. Así será como entregará los sobres de tratamiento a la psiquiatra tratante, entonces ésta será ciega al tratamiento ya que sólo manejará los sobres con el número del paciente, sin saber a qué grupo de tratamiento pertenece cada uno de ellos. Además, tal como se explicó en el punto de "tratamientos a administrar", tanto la NAC como el placebo vendrán en la misma presentación farmacéutica, con lo cual los pacientes también serán ciegos a la farmacoterapia recibida.
- d. Administración del Tratamiento: Previo a la administración del tratamiento, se tomará a cada paciente un test para la detección de drogas en orina y un examen sanguíneo basal que incluya hemograma, glicemia, pruebas hepáticas y creatininemia, entre otros. Posteriormente el médico o enfermero(a) del equipo investigador entregarán los sobres con la farmacoterapia a administrar a cada paciente, en el centro de tratamiento correspondiente. Inicialmente el médico o





enfermero(a) supervisará la ingesta del fármaco y solicitará al paciente permanecer en la unidad clínica por dos horas, período en el cual se registrará si existe alguna RAM inmediata y se le controlará la presión arterial, frecuencia cardíaca y temperatura corporal. Será el paciente el responsable de la ingesta de las siguientes dosis de medicamentos y de informar acerca de posibles RAM que surjan antes del control siguiente, una vez que se retire del centro de atención.

- e. Controles en los Centros de Atención Clínica: se le pedirá a cada paciente que asista dos veces por semana a su centro de tratamiento, durante las cuatro semanas que dura el estudio. En cada visita del paciente se evaluarán distintos parámetros, los que se describirán posteriormente en esta sección del proyecto. Además en cada visita el paciente recibirá una intervención de tipo psicoeducativa, consejería u ocupacional, según el protocolo de atención del centro de tratamiento donde se esté realizando el estudio. No recibirá psicoterapia propiamente tal como tratamiento.
- f. Evaluación del Cumplimiento Terapéutico: Para esto se consultará a los pacientes acerca de la toma de sus medicamentos y de las dificultades que pudiesen haber tenido con ello, en cada visita al centro de tratamiento. Para evaluar el grado de veracidad de esta información, se aplicará a cada paciente el Test de Morisky-Green semanalmente, en sus visitas de control.
- g. Evaluación de Tolerabilidad: ésta se evaluará consultando a los pacientes acerca de las posibles reacciones adversas a los medicamentos (RAM) administrados, las cuales serán registradas en la ficha de control en cada visita y, al mismo tiempo, se evaluará consignando cada vez que un paciente abandone el tratamiento a causa de éstas.
- h. Evaluación de Seguridad: ésta se evaluará consignando las posibles RAM graves que surgieran tras la administración de alguno de los tratamientos. En dicho caso se activará el protocolo de seguridad correspondiente, normado por el ISP de Chile<sup>71</sup>, otorgando al paciente todas las atenciones médicas necesarias para proteger su vida e integridad física y mental. Así mismo se notificará de inmediato acerca de este evento al Comité de Farmaco-Vigilancia y al Comité de Ética del servicio correspondiente.
- i. Evaluación del Tiempo de Abstinencia: se medirá registrando en la ficha clínica los días sin consumo de PBC reportados por el paciente y a través de la aplicación de test de drogas en orina los que se realizarán semanalmente a éstos, en sus visitas de control a los centros de atención correspondientes.
- j. Evaluación de los Síntomas de Abstinencia: Para ello se registrarán en la ficha clínica de cada paciente, los síntomas que ellos refieran espontáneamente como molestias tras cesar el consumo de PBC. En conjunto con esto se les aplicará, tanto al ingreso como en cada visita al centro de atención clínica, el CSSA, cuestionario de abstinencia de cocaína previamente descrito y validado al español recientemente.

k. Evaluación del Craving: El mismo día del ingreso al estudio se solicitará a cada paciente que informe, en la escala Escala Visual Análoga previamente descrita (EVA, de 1 a 100), cuál era su apetencia por el consumo de PBC en la semana previa al







ingreso y cuál es ésta al momento de la consulta. En paralelo se les aplicará la escala de *craving* de cocaína CCQ-N-10, también ya descrita y validada al español recientemente.

## H. ANÁLISIS ESTADÍSTICO:

El resultado principal de este ensayo se describirá como sigue:

- la proporción de pacientes que estuvo de acuerdo para entrar en el ensayo,
- · las diferencias entre aquellos que entraron y aquellos que rehusaron,
- · las características de la muestra,
- la adhesión al tratamiento, y
- el número y las características de los abandonos durante el seguimiento.

Se compararán las características de los participantes en cada brazo del ensayo. Las variables a comparar serán sexo, edad, comorbilidad, tiempo de consumo de PBC, severidad del trastorno por uso de PBC y *craving* basal por PBC, para verificar la homogeneidad entre los grupos.

- Se compararán los resultados primarios en el seguimiento a las cuatro semanas, a saber: craving y duración media de los días de abstinencia de PBC.
- Después de verificar la distribución del *craving y* la duración media de los días de abstinencia de PBC en ambos grupos, se analizará un modelo ajustando de acuerdo a la severidad del trastorno por uso de PBC en la línea base, dado que ésta es la variable más relevante reportada en la literatura que pudiese influir en la abstinencia.
- Las diferencias en el resultado primario por grupo (con el ajuste por severidad) serán reportados junto con sus intervalos de confianza del 95%.

Los resultados serán analizados utilizando el programa estadístico SPSS y R. De acuerdo a las variables de resultado a evaluar, los análisis serán:

- Para evaluación del Craving: se analizará aplicando pruebas de comparación de medias (T Student, bajo normalidad verificada con Kolmogorov Smirnov, o U Mann Whitney, en caso contrario) para muestras independientes, considerando las mediciones iniciales (antes de que se aprecie mucha deserción).
- Para evaluación del tiempo de abstinencia de PBC: Se compararán los días de abstinencia mediante un análisis de supervivencia con el estimador de Kaplan-Mier. En caso de encontrar aumento siginificativo de los días de abstinencia de PBC en el grupo de tratamiento con NAC se hará un estudio de correlación (Pearson, si se verifica normalidad; Spearman en caso contrario) entre las variables cuantitativas medidas a los individuos y días de abstinencia.
- Para evaluación de la tasa de caídas en el consumo de PBC: Se compararán las tasas de caídas en el consumo de PBC mediante un modelo lineal generalizado mixto, con respuesta Poisson y tiempos entre recaídas exponencial. En caso de sobre-dispersión, se considerará un modelo con respuesta Binomial Negativa.







Se realizará comparación de medias entre grupos experimental y control mediante ANOVA de medidas repetidas (si se verifica normalidad con Kolmogorov Smirnov y homocedasticidad con Fisher) o análisis tipo ANOVA no paramétrico para medidas repetidas (en caso contrario). Además es importante mencionar que los datos incompletos por abandono del estudio, ya sea que exista o no retorno, deberán ser considerados para los análisis.

# I. RESULTADOS ESPERADOS DE LA INVESTIGACIÓN

Se espera que, gracias a la utilización de la NAC, los pacientes con dependencia de PBC ingresados al estudio reduzcan significativamete su urgencia por consumir dicha sustancia y prolonguen el tiempo de abstinencia de la misma. Por otra parte se espera que gracias a la NAC estos pacientes reduzcan sus caídas en el consumo de PBC y que, gracias a su observación sistemática, se pueda conocer de mejor manera el cuadro clínico del síndrome de abstinencia de PBC y contar con un instrumento de medición de éste. Finalmente se espera que durante este estudio se logre capacitar a equipos multidisciplinarios que trabajen con pacientes dependientes de PBC en la provincia de Concepción para mejorar parte del proceso diagnóstico y terapéutico en cada uno de sus centros de atención clínica.

# 5. CONSENTIMIENTO INFORMADO Y ASPECTOS ÉTICOS:

Los clínicos participantes de este estudio informarán al paciente sobre la naturaleza del proyecto y solicitaran su participación voluntaria junto a la autorización explícita para obtener información sobre el tratamiento recibido desde su ficha clínica. Aquellos que acepten participar deberán firmar un consentimiento informado previo a su inclusión en el estudio. El modelo de Consentimiento Informado se basa en los requerimientos del Ministerio de Salud y del Instituto de Salud Pública de Chile y deberá ser aprobado por los Comités de Ética de los respectivos Servicios de Salud a los que los pacientes se encuentren adscritos, así como por el Comité de Ética de la Facultad de Medicina de la Universidad de Concepción.

Los aspectos éticos de este proyecto de investigación dicen relación con que se trata de una investigación en seres humanos a los cuales se les administrarán, aleatoriamente y de modo ciego, dos tratamientos distintos: uno biológicamente activo que, dada la evidencia científica internacional existente a la fecha, se espera sea efectivo para reducir el *craving* de PBC y el otro, consistente en una formulación farmacéutica biológicamente inactiva, conocida como placebo, que por lo mismo probablemente no es efectiva para tratar el síntoma en el que se focaliza esta investigación.

Respecto de este último punto cabe destacar que, ateniéndose a los principios éticos para las investigaciones médicas en seres humanos contenidos en la Declaración de Helsinki de la Asociación Médica Mundial<sup>71</sup>, es factible realizar una investigación con placebo siempre y cuando no se cuente con una terapia probada y existente, que es lo que ocurre en







Chile (y en el mundo) con el caso del manejo de la dependencia y del síndrome de abstinencia de la PBC.

Por otro lado, el fármaco a utilizar, cual es la N-Acetilcisteína (NAC), además de reunir evidencia científica acerca de su utilidad en pacientes con trastornos por consumo de cocaína y otras drogas, es un fármaco ya conocido en Chile desde hace años, utilizado con diversos fines, en dosis superiores a las que se usarían en este estudio y es muy seguro de utilizar.

En relación con todo lo anterior, en este proyecto se adjunta una carta en la cual la investigadora responsable del mismo declara que sus actuaciones están en pleno acuerdo con:

- la Declaración de Helsinki en todas sus versiones,
- con las normas de Buenas Prácticas Clínicas (GCP) establecidas por la Organización Mundial de la Salud,
- con las Normas Éticas Internacionales para las investigaciones biomédicas con sujetos humanos (Organización Panamericana de la Salud y por el Consejo de Organizaciones Internacionales de las Ciencias Médicas,
- con las Directrices Operativas para los Comités de Ética en Investigación Biomédica y
- con las Regulaciones Nacionales:
  - o LEY Nº 19.628 sobre "Protección de la vida privada o protección de datos de carácter personal", Publicada en el Diario Oficial de 28 de agosto de 1999,
  - Norma Técnica N° 57 del 04 de Junio del 2001, del Ministerio de Salud del Gobierno de Chile, Regulación de la Ejecución de Ensayos Clínicos que utilizan Productos Farmacéuticos en Seres Humanos<sup>72</sup>;
  - Ley Nº 20120 y su Reglamento sobre "La Investigación Científica en el Ser Humano, Su Genoma, y Prohíbe la Clonación Humana" con vigencia desde el 22.09.2006,
  - Decreto N°114 promulgado el 22.11.2010, que aprueba su Reglamento, Decreto 30 promulgado el 05.07.2012, que modifica dicho reglamento y
  - o la Ley 20.584, de título "Regula los derechos y deberes que tienen las personas en relación con acciones vinculadas a su atención en salud", promulgada el 13-04-2012 y en vigencia desde el 01.10.2012.

Se adjunta también la carta de presentación de este proyecto al Comité de Ética de la Universidad de Concepción, así como el consentimiento informado que deberán firmar los pacientes que acepten ingresar al estudio, el cual en caso de ser revocado no afectará la relación médico-paciente ni perjudicará de ningún modo a este último.

En cuanto a lo que dice relación con el manejo de muestras biológicas, es importante aclarar que los exámenes que serán realizados a los pacientes que ingresen al estudio, son exámenes que se hacen rutinariamente al ingreso de estos a sus centros de atención en salud mental, por el personal de salud que allí trabaja, el cual se encuentra debidamente capacitado









y acreditado para estos efectos, quienes además adscriben a la normativa nacional vigente de bioseguridad relacionada con el manejo de muestras biológicas.

Por otra parte, respecto de la duración de la intervención y los posibles riesgos o pérdida de posibilidad de otra intervención para el paciente en el mismo período, es importante destacar que en el manejo general de los pacientes con dependencia de drogas, ingresados a los centros de salud mental en convenio SENDA-MINSAL, las primeras cuatro semanas de atención de estos, están dedicadas básicamente a la evaluación bio-psico-social del paciente, así como a reforzar su motivación a tratamiento y es justamente en ese período en el cual, muchas veces por no contar con las herramientas farmacológicas adecuadas para el manejo de los síntomas de abstinencia, existe la mayor tasa de abandono del proceso. Es en ese contexto entonces, que se propone en este estudio iniciar precozmente la farmacoterapia, de modo de facilitar, entre otras cosas, la adherencia al proceso de evaluación e ingreso al centro.

Finalmente y para cerrar este punto, es relevante mencionar que este proyecto cautela que el protocolo de intervención adscriba plenamente a los puntos básicos que debe resguardar toda investigación médica, tales como "...proteger la vida, la salud, la intimidad y la dignidad del ser humano...apoyarse en un profundo conocimiento de la bibliografía científica...ser llevada a cabo por personas científicamente calificadas y bajo la supervisión de un médico clínicamente competente...ser precedida de una cuidadosa comparación de los riesgos calculados con los beneficios previsibles...tener la posibilidad de suspender el experimento en marcha si se observa que los riesgos son más importantes que el beneficio..." y que los "...participantes sean voluntarios e informados...", entre otros.

# 6. DOCUMENTACIÓN DEL CONSENTIMIENTO INFORMADO:

Se anexa junto a la documentación entregada al Comité Ético Científico al momento de presentar este proyecto.

#### REFERENCIAS

- 1. Toffoli F, Avico U. Coca paste: Residues from the industrial extraction of cocaine ecgonine and anhydroecgonine. *Bulletin of Narcotics* 1965; 17 (4): 27 -36.
- Pascale A, Hynes M, Cumsille F, Bares C. Consumo de pasta base de cocaína en América del Sur: revisión de los aspectos epidemiológicos y médico-toxicológicos. Inter-American Drug Abuse Control Commission Inter-American Observatory on Drugs: Organización de los Estados Americanos (OEA); 2014.
- 3. Prieto JP, Scorza MC. Pasta Base de Cocaína. Uruguay: Laboratorio de Biología Celular, Instituto de Investigaciones Biológicas Clemente Estable; 2010.
- 4. Maass J, Kirberg A. La epidemia de cocaína: morbo en el norte de Chile. Revista de Psiquiatría. 1990; 7: 639-647.







- 5. Comisión interamericana para el control del abuso de drogas, CICAD. Informe del Uso de Drogas en las Américas 2015. Washington, DC: Organización de los Estados Americanos, 2015.
- Servicio Nacional Para la Prevención y Rehabilitación Del Consumo De Drogas y Alcohol, SENDA. Décimo Primer Estudio Nacional de Drogas en Población General de Chile, 2014. Santiago de Chile: Ministerio del Interior y Seguridad Pública. Gobierno de Chile. 2015.
- Pérez J. Clínica de la adicción a pasta base de cocaína. Rev Chil Neuro-psiquiatr 2003;
   55-63.
- 8. Iraugi Castillo I., Corcuera Bilbao N. Craving: concepto, medición y terapéutica. Norte De Salud Mental. 2008;32(1): 9-22.
- 9. Chesa Vela D, Abadías ME, Fernández Vidal E, Izquierdo Munuera E, Sitjas Carvacho M. El craving, un componente esencial en la abstinencia. Rev. Asoc. Esp. Neuropsiq. 2004; 89: 93-112.
- 10. World Health Organization, WHO. Global Burden. (Online). Disponible en: http://www.who.int/substance\_abuse/facts/global\_burden/en/ [Accessed 16 Febrero 2016].
- 11. World Health Organization, WHO. Global Burden. (Online). Disponible en: http://www.who.int/substance\_abuse/facts/global\_burden/en/ [Accessed 16 Febrero 2016].
- 12. Oficina de las Naciones Unidas Contra la Droga y el Delito (UNODC). Informe Mundial sobre las Drogas 2015. Resumen Ejecutivo. *Naciones Unidas ed.* Nueva York. 2015.
- 13. Degenhardt L, Whiteford HA, Ferrari AJ, Baxter AJ, Charlson FJ, Hall WD, et als. Global burden of disease attributable to illicit drug use and dependence: findings from the Global Burden of Disease Study 2010. Lancet. 2013: 9; 382(9904):1564-74.
- 14. Servicio Nacional de Drogas y Alcohol, SENDA. Área de Tratamiento y Rehabilitación: Informe Semestral 2015 Evaluación Técnica Convenio. [Online]. Disponible en: http://www.senda.gob.cl/media/2015/06/PDF-453-KB-Planes-Tto.-Personas.pdf [Accedido 16 Febrero 2016]
- 15. Asociación Americana de Psiquiatría, APA. Guía de Consulta de los Criterios Diagnósticos del DSM-5 (1st ed.) Washington, DC: American Psychiatric Publishing, 2014.
- 16. Regier D, Farmer M, Rae D, Locke B, Keith S, Judd L, et al. Co-morbidity of mental disorders with alcohol and other drug abuse: results from the epidemiologic catchment area (ECA) study. *JAMA*. 1990: 264(19);2511-8.
- 17. Vergara-Moragues E, González-Saiz F, Lozano OM, Betanzos Espinosa P, Fernández Calderón F, Bilbao-Acebos I, Pérez García M, Verdejo García A. Psychiatric comorbidity in cocaine users treated in therapeutic community: substance-induced versus independent disorders. Psychiatry Res. 2012;200(2-3):734-41.







- 18. Zubaran C, Foresti K, Thorell MR, Franceschini PR. Anxiety symptoms in crack cocaine and inhalant users admitted to a psychiatric hospital in southern Brazil. Rev Assoc Med Bras. 2013;59(4):360-7.
- 19. Araos P, Vergara-Moragues E, Pedraz M, Pavón FJ, Campos Cloute R, Calado M, Ruiz JJ, García-Marchena N, et al. Psychopathological comorbidity in cocaine users in outpatient treatment. Adicciones. 2014;26(1):15-26.
- 20. Benedict ES, Gorman A, van Gorp W, Foltin RW, Vadhan NP. Self-reported attention and mood symptoms in cocaine abusers: relationship to neurocognitive performance. Psychiatry Res. 2014;219(3):598-603.
- 21. Roy É, Jutras-Aswad D, Bertrand K, Dufour M, Perreault M, Laverdière É, Bene-Tchaleu F, Bruneau J. Anxiety, mood disorders and injection risk behaviors among cocaine users: Results from the COSMO study. Am J Addict. 2015;24(7):654-60.
- 22. Herrero MJ, Domingo-Salvany A, Torrens M, Brugal MT. Psychiatric comorbidity in young cocaine users: induced versus independent disorders. *Addiction*. 2007: 103(2); 284-293.
- 23. Restrepo CS, Carrillo JA, Martínez S, Ojeda P, Rivera AL, Hatta A. Pulmonary Complications from Cocaine and Cocaine-based Substances: Imaging Manifestations. *Radiographics*. 2007: 27(4); 941-956.
- 24. Mançano A, Marchiori E, Zanetti G, Escuissato DL, Duarte BC, Apolinário Lde A. Pulmonary complications of crack cocaine use: high-resolution computed tomography of the chest. J Bras Pneumol. 2008; 34(5):323-7.
- 25. Story A, Bothamley G, Hayward A. Crack cocaine and infectious tuberculosis. Emerg Infect Dis. 2008:14(9);1466-9.
- 26. Drent M, Wijnen P, Bast A. Interstitial lung damage due to cocaine abuse: pathogenesis, pharmacogenomics and therapy. Curr Med Chem. 2012;19(33):5607-11.
- 27. Leece P, Rajaram N, Woolhouse S, Millson M. Acute and chronic respiratory symptoms among primary care patients who smoke crack cocaine. J Urban Health. 2013;90(3):542-51.
- 28. Haim DY, Lippmann ML, Goldberg SK, Walkenstein MD. The pulmonary complications of crack cocaine: a comprehensive review. CHEST Journal. 1995: 107(1); 233-240.
- 29. Pascale A, Negrín A, Ormaechea R. Estudio preliminar de la repercusión pulmonar por consumo de pasta base de cocaína. Arch Bronconeumol. 2011: 47(2);108.
- 30. Santis R, Hidalgo CG, Hayden V, Anselmo E, Rodríguez J, Dreyse J, et al. Consumo de sustancias y conductas de riesgo en consumidores de pasta base de cacaína no consultantes a servicios de rehabilitación. Rev Méd Chile. 2007: 135(1); 45-53.
- 31. Valenzuela E, Larroulet P. La relación droga y delito. *Estudios públicos*. 2010: 119; 33-62.
- 32. Servicio nacional para la prevención y rehabilitación del consumo de drogas y alcohol, SENDA. Variables asociadas a la necesidad y asistencia a tratamiento en personas con trastornos por consumo de drogas y alcohol en Chile. [Online]. Disponible en Versión 2. Fecha: 20 de marzo de 2017







http://www.senda.gob.cl/media/boletines/Boletin%2021%20Variables%20asociadas%20a%20la%20necesidad%20y%20asistencia%20a%20tratamiento%20en%20personas%20con%20trastornos%20por%20consumo%20de%20drogas%20y%20alcohol%20en%20Chile.pdf (Accedido 16 febrero 2016).

- 33. Servicio Nacional Para la Prevención y Rehabilitación Del Consumo De Drogas y Alcohol, SENDA. Tratamiento. Disponible en: http://www.senda.gob.cl/tratamiento/presentacion/ (Accedido 17 febrero 2016).
- 34. Quintero GC. Role of nucleus accumbens glutamatergic plasticity in drug addiction. Neuropsychiatric Disease and Treatment. 2013: 9; 1499–1512.
- 35. Asevedo E, Mendes AC, Berk M, Brietzke E. Systematic review of N-acetylcysteine in the treatment of addictions. *Revista Brasileira de Psiquiatria*. 2014: 36(2); 168-175.
- 36. Baker DA, McFarland K, Lake RW, Shen H, Tang XC, Toda S, et al. Neuroadaptations in cystine-glutamate exchange underlie cocaine relapse. *Nat Neurosci.* 2003: 6;743-749.
- 37. LaRowe SD, Mardikian P, Malcolm R, Myrick H, Kalivas P, McFarland K at al. Safety and tolerability of N-acetylcysteine in cocaine-dependent individuals. *American Journal on Addictions*. 2006: 15(1), 105-110.
- 38. Mardikian PN, LaRowe SD, Hedden S, Kalivas PW, Malcolm RJ. An open-label trial of N-acetylcysteine for the treatment of cocaine dependence: a pilot study. *Prog Neuropsychopharmacol Biol Psychiatry*. 2007: 31; 389-394.
- 39. LaRowe SD, Kalivas PW, Nicholas JS, Randall PK, Mardikian PN, Malcolm RJ. A double-blind placebo-controlled trial of N-acetylcysteine in the treatment of cocaine dependence. Am J Addict. 2013: 22(5); 443-52
- 40. LaRowe SD, Myrick H, Hedden S, Mardikian P, Saladin M, McRae A, et al. Is cocaine desire reduced by N-acetylcysteine? *Am J Psychiatry*. 2007: 164;1115-1117.
- 41. Amen SL, Piacentine LB, Ahmad ME, Li SJ, Mantsch JR, Risinger RC, et al. Repeated N-acetyl cysteine reduces cocaine seeking in rodents and craving in cocaine-dependent humans. *Neuropsychopharmacology*. 2011: 36(4); 871-878.
- 42. Kupchik YM, Moussawi K, Tang XC, Wang X, Kalivas BC, Kolokithas R, et al. The effect of N-acetylcysteine in the nucleus accumbens on neurotransmission and relapse to cocaine. *Biological psychiatry*. 2012: 71(11), 978-986.
- 43. McClure EA, Gipson CD, Malcolm RJ, Kalivas PW, Gray KM. Potential role of Nacetylcysteine in the management of substance use disorders. CNS drugs. 2014: 28(2); 95-106.
- 44. Deepmala, Slattery J, Kumar N, Delhey L, Berk M, Dean O, et al. Clinical trials of Nacetylcysteine in psychiatry and neurology: A systematic review. Neurosci Biobehav Rev. 2015: 55;294-321.
- 45. Brahm J, Silva G, Palma R. Paracetamol overdose: a new form of suicide in Chile and the value of N-acetylcysteine administration. *Revista medica de Chile*. 1992: 120(4); 427-429.







- 46. Instituto de Salud Pública (ISP), Ministerio de Salud (MINSAL), Gobierno De Chile. Sistema de Consultas de Productos Registrados. [Online]. Disponible en: http://registrosanitario.ispch.gob.cl/ (Accedido el 16 Febrero 2016).
- 47. Sociedad Iberoamericana de Información Científica. Colección de trabajos Claves. Actualizan el Uso Terapéutico de la N-Acetilcisteína y los Mecanismos de Acción Involucrados. (Online) Disponible en: https://www.siicsalud.com/pdf/tc\_acetilcisteina\_22513.pdf. (Accedido el 16 Febrero 2016)
- 48. Camí J., Farré M. (2003). Drug Addiction. N Engl J Med; 349:975-986.
- 49. Koob GF. (1992) Drugs of abuse: anatomy, pharmacology and function of reward pathways. Trends Pharmachol Sci; 13:177-184.
- 50. Cornish JL, Duffy P, Kalivas PW (1999). A role for nucleus accumbens glutamate transmission in the relapse to cocaine- seeking behavior. *Neurosci.* 93:1359-1367.
- 51. Tzschentke TM, Schmidt WJ. Glutamatergic mechanisms in addiction. *Mol Psychiatry*. 2003: 8; 373-82.
- 52. Uys JD, LaLumiere RT. Glutamate: the new frontier in pharmacotherapy for cocaine addiction. CNS Neurol Disord Drug Targets. 2008: 7; 482-491.
- 53. Martinez-Raga J, Knecht C, Ramírez N, Szerman N. Sistemas de neurotransmisión glutamatérgica y adicción a la cocaína. Progresos en el tratamiento farmacológico. *Rev Psiquiatr Urug 2009;73(1):63-72*.
- 54. Gass JT, Olive MF. Glutamatergic substrates of drug addiction and alcoholism. Biochem Pharmacol 2008; 75:218-265.
- 55. López Durán A., Becoña Iglesias E. El craving en personas dependientes de la cocaína. Anales de psicología. 2006; 22(2): 205-211.
- 56. Gawin F, Kleber H. Envolving Conceptualizations of Cocaine Dependence. The Yale Journal of Biology and Medicine. 1988: 61; 123-136.
- 57. Halikas, J.A, Kuhn, K.L., Crosby, R., Carlson, G. y Crea, F. The measurement of *craving* in cocaine patients using the Minnesota cocaine craving scale. *Comprehensive Psychiatry.* 1991; 32: 22-27.
- 58. Iraurgi Castillo I, Trujols Albet J, Jiménez-Lerma JM, Landabaso M. Reliability and validity of the Spanish adaptation of the brief form of the Cocaine Craving Questionnaire-Now (CCQ-N-10). *Adicciones*. 2009;21(3):195-202.
- 59. Tiffany, S.T., Singlenton, E., Haertzen, C.A. y Henningfield, I.E. The development of a cocaine craving questionnaire. Drug and Alcohol Dependence. 1993; 34: 19-28.
- 60. Tejero, A., Trujols, J. y Siñol, N. Evaluación del craving de cocaína. En: J. Pérez de los Cobos, A. Tejero y J. Trujols, *Instrumentos clínicos para la evaluación de la dependencia de la cocaína*. 2003: 23-50.
- 61. Kampman KM, Volpicelli JR, McGinnis DE, Alterman AI, Weinrieb RM, D'Angelo L, Epperson LE. Reliability and validity of the Cocaine Selective Severity Assessment Addict Behav. 1998;23(4):449-61.







- 62. Pérez de los Cobos J, Trujols J, Siñol N, Vasconcelos e Rego L, Iraurgi I, Batlle F. Psychometric properties of the Spanish version of the Cocaine Selective Severity Assessment to evaluate cocaine withdrawal in treatment-seeking individuals. *J Subst Abuse Treat.* 2014;47(3):189-96.
- 63. Kampman KM, Lynch KG, Pettinati HM, Spratt K, Wierzbicki MR, Dackis C, O'Brien CP. A double blind, placebo controlled trial of modafinil for the treatment of cocaine dependence without co-morbid alcohol dependence. *Drug Alcohol Depend.* 2015: 1;155:105-10.
- 64. Ahmadi J, Kampman KM, Oslin DM, Pettinati HM, Dackis C, Sparkman T. Predictors of treatment outcome in outpatient cocaine and alcohol dependence treatment. Am J Addict. 2009 Jan-Feb; 18(1):81-6.
- 65. Consejo Nacional para el Control de Estupefacientes (CONACE). Orientaciones Técnicas Tratamiento del consumo problemático de alcohol y drogas y otros trastornos de salud mental en adolescentes infractores de ley. Santiago, *Ministerio del Interior y Seguridad Pública. Gobierno de Chile.* 2007.
- 66. Servicio Nacional Para la Prevención y Rehabilitación Del Consumo De Drogas y Alcohol, SENDA. Normas y Orientaciones Técnicas de los Planes de Tratamiento y Rehabilitación para Personas Adultas con Problemas Derivados del Consumo de Drogas. Convenio SENDA-MINSAL 2012. Santiago, Ministerio del Interior y Seguridad Pública. Gobierno de Chile. 2012.
- 67. Ministerio de Salud (MINSAL). Guía Clínica AUGE "Consumo perjudicial y Dependencia de alcohol y otras drogas en personas menores de 20 años". Santiago: MINSAL, 2013.
- 68. Ferrando, L Bobes J, Gibert J. MINI International Neuropsychiatric Interview. Versión en Español 5.0.0 DSM-IV. Barcelona, España. 2000.
- 69. Bobes J, Portilla M, Bascarán M, Sáiz P, Bousoño M. Banco de Instrumentos Básicos para la Práctica de la Psiquiatría Clínica. (3ª Ed.) Barcelona: Psiquiatría Editores SI. 2004.
- 70. Rodríguez Chamorro MA, García-Jiménez E, Amarilesc P, Rodríguez Chamorro A, Fause MJ. Revisión de tests de medición del cumplimiento terapéutico utilizados en la práctica clínica. *Aten Primaria*. 2008;40(8):413-7
- 71. Asociación Médica Mundial. Declaración De Helsinki. (Online) Disponible en: http://www.conicyt.cl/fondecyt/files/2012/10/Declaraci%C3%B3n-de-Helsinki-de-la-Asociaci%C3%B3n-M%C3%A9dica-Mundial.pdf (Accedido 27 junio 2016).
- 72. Ministerio de Salud del Gobierno de Chile, Instituto de Salud Pública. Norma Técnica N° 57: Regulación de la Ejecución de Ensayos Clínicos que Utilizan Productos Farmacéuticos en Seres Humanos. Santiago de Chile, 2001.









#### **ANEXOS**

#### 1. FLUJOGRAMA Y PLAN DE TRABAJO:

#### a) Flujograma:



Versión 2. Fecha: 20 de marzo de 2017









## b) Plan de trabajo:

| ETAPAS Y/O ACTIVIDADES | PRIMER AÑO DE INVESTIGACIÓN trimestres | | | | SEGUNDO AÑO DE INVESTIGACIÓN trimestres | | | |
|---|---|---|---|---|---|---|---|---|
| | Envio solicitud aprobación a comités de ética correspondientes | X | | | | | | |
| Organización del equipo de trabajo | X | | | | | | | |
| Coordinación con centros de atención de pacientes con drogodependencias | X | | | | | | | |
| Confección de cuestionario para recogida de datos sociodemográficos y clínicos | X | | | | | | | |
| Selección de entrevistadores y tratantes | X | | | | | | | |
| Capacitación de entrevistadores y tratantes | X | | | | | | | |
| Entrevistas a usuarios | | X | X | X | | | | |
| Selección de la muestra | | X | X | X | | | | |
| Recolección datos clínicos | | X | X | X | | | | |
| Procesamiento de datos en busca de índices de validez del instrumento de medida de craving | | X | X | X | | | | |
| Aplicación Tratamiento a Pacientes | | | X | X | X | X | | |
| Evaluación de tratamientos | | | X | X | X | X | | |
| Procesamiento de datos acerca de resultados de tratamientos | | | | | X | X | X | |
| Análisis de datos | | | | | X | X | X | |
| Publicación de resultados | | | | | 1 | | | X |

